CLINICAL TRIAL: NCT06661564
Title: Identification de Biomarqueurs Diagnostiques Dans Les Larmes de Patients Atteints de Maladie d'Alzheimer : l'étude Pilote COG-EYE
Brief Title: Identification of Diagnosis Biomarkers in the Tears of Alzheimer's Disease Patients: The COG-EYE Pilot Study
Acronym: COG-EYE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DR240140
Record Dates: First submitted 2024-10-16; First posted 2024-10-28 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Disease
Keywords: biomarkers; tears; metabolomic; lipidomic; Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease; Lacerations | interventions — tau Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients with AD dementia (Active Comparator): Patient ≥ 18 years old with AD at a major stage according to the 2018 NIA-AA criteria (dementia)
  Interventions: Other: Basal tear collection for the analysis of metabo-lipidomic profiles and concentrations of protein biomarkers (Tau, phosphorylated Tau, Aβ 1-40, and Aβ 1-42)
- Patients with AD Mild Cognitive Impaiment (MCI) (Active Comparator): Patient ≥ 18 years old with AD at a minor stage according to the 2018 NIA-AA criteria (Mild Cognitive Impairment)
  Interventions: Other: Basal tear collection for the analysis of metabo-lipidomic profiles and concentrations of protein biomarkers (Tau, phosphorylated Tau, Aβ 1-40, and Aβ 1-42); Other: Collection of a blood sample (5 mL) for blood biomarkers analysis
- Healthy controls (Sham Comparator): Participants ≥ 18 years old with no known central neurological pathology, no cognitive decline, and matched by age (± 2 years) and sex with a patient from AD-MCI group
  Interventions: Other: Basal tear collection for the analysis of metabo-lipidomic profiles and concentrations of protein biomarkers (Tau, phosphorylated Tau, Aβ 1-40, and Aβ 1-42)

INTERVENTIONS:
Other: Basal tear collection for the analysis of metabo-lipidomic profiles and concentrations of protein biomarkers (Tau, phosphorylated Tau, Aβ 1-40, and Aβ 1-42) — Collection of a tear volume of (i) 2 x 5µL using glass microcapillary tubes and (ii) 12µL using Schirmer strips after the instillation of anesthetic eye drops for metabo-lipidomic analysis and multiplexing of protein markers
Other: Collection of a blood sample (5 mL) for blood biomarkers analysis — Collection of a blood sample (5 mL) for blood biomarkers analysis.
  Arms: Patients with AD Mild Cognitive Impaiment (MCI)

SUMMARY:
The diagnosis of Alzheimer's disease (AD) relies on the detection of protein biomarkers, particularly in cerebrospinal fluid (e.g., Aβ and phosphorylated Tau) or through brain imaging. The invasive nature of lumbar puncture and the numerous contraindications have driven the search for early and reliable diagnostic biomarkers for AD.

Human tears are an accessible biological fluid that has proven relevant in the biomarker search strategy for both ophthalmological and systemic diseases, especially neurodegenerative conditions. Advances in methods for low-volume analysis have facilitated the identification of tear biomarkers. Total tau has been reported as elevated in the tears of patients with AD compared to controls (n=65). Additionally, metabo-lipidomic analyses offer several advantages (accessibility, non-invasiveness, reproducibility) and also appear promising as a diagnostic tool for systemic and neurodegenerative diseases, such as amyotrophic lateral sclerosis. This supports the relevance of comparing both AD proteins biomarkers and metabo-lipidomic signatures in the tears of patients with AD (Mild Cognitive Impairement (MCI) and dementia) with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Participant affiliated in French Social Security scheme
* Informed and written consent from the participant

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Participant under judicial protection measures
* Participant under guardianship or curatorship
* Contraindications to participation in the research:

Other neurodegenerative disease Any eye drops or treatment that may interfere with tear production Occasional or permanent contact lens use within the last 3 months Eye surgery ≤3 months Any ocular pathology other than refractive errors, oculomotor disorders, amblyopia Any general pathology other than AD with ocular implications

-Inability to perform tear collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Concentration of total Tau proteins in basal tears of patients with AD vs healthy volunteers | At inclusion
  12μL of tears will be collected using Schirmer strips after instillation of an anaesthetic eye drop. A multiplex analysis for the detection of protein of interest
Concentration of phosphorylated Tau proteins in basal tears of patients with AD vs healthy volunteers | At inclusion
  12μL of tears will be collected using Schirmer strips after instillation of an anaesthetic eye drop. A multiplex analysis for the detection of protein of interest
Concentration of Amyloid β 1-40 proteins in basal tears of patients with AD vs healthy volunteers | At inclusion
  12μL of tears will be collected using Schirmer strips after instillation of an anaesthetic eye drop. A multiplex analysis for the detection of protein of interest
Concentration of Amyloid β 1-42 in basal tears of patients with AD vs healthy volunteers | At inclusion
  12μL of tears will be collected using Schirmer strips after instillation of an anaesthetic eye drop. A multiplex analysis for the detection of protein of interest
Lipids in basal tears of patients with AD vs healthy volunteers | At inclusion
  Collection of tears (5μL) using a glass micropipette without local anaesthetic. Lipids in tears of patients with AD vs healthy volunteers
Metabolites in basal tears of patients with AD vs healthy volunteers | At inclusion
  Collection of tears (5μL) using a glass micropipette without local anaesthetic. Metabolites in tears of patients with AD vs healthy volunteers

SECONDARY OUTCOMES:
Concentration of total Tau proteins in tears vs plasma and Cerebral spinal fluid (CSF) within patients with AD-MCI | At inclusion
  12μL of tears will be collected using Schirmer strips after instillation of an anaesthetic eye drop. A multiplex analysis for the detection of protein of interest
Concentration of phosphylated Tau proteins in tears vs plasma and Cerebral spinal fluid (CSF) within patients with AD-MCI | A inclusion
  12μL of tears will be collected using Schirmer strips after instillation of an anaesthetic eye drop. A multiplex analysis for the detection of protein of interest
Concentration of Amyloid β 1-40 proteins in tears vs plasma and Cerebral spinal fluid (CSF) within patients with AD-MCI | A inclusion
  12μL of tears will be collected using Schirmer strips after instillation of an anaesthetic eye drop. A multiplex analysis for the detection of protein of interest
Concentration of Amyloid β 1-42 proteins in tears vs plasma and Cerebral spinal fluid (CSF) within patients with AD-MCI | A inclusion
  12μL of tears will be collected using Schirmer strips after instillation of an anaesthetic eye drop. A multiplex analysis for the detection of protein of interest
Lipids in tears vs plasma and Cerebral spinal fluid (CSF) within patients with AD-MCI | At inclusion
  Collection of tears (5μL) using a glass micropipette without local anaesthetic. Identification of lipids in basal tears using liquid chromatography-mass spectrometry.
Metabolites in tears vs plasma and Cerebral spinal fluid (CSF) within patients with AD-MCI | At inclusion
  Collection of tears (5μL) using a glass micropipette without local anaesthetic. Identification of metabolites in basal tears using liquid chromatography-mass spectrometry.
Concentration of total Tau proteins in basal tears of patients with AD-dementia vs patients with AD-MCI | At inclusion
  12μL of tears will be collected using Schirmer strips after instillation of an anaesthetic eye drop. A multiplex analysis for the detection of protein of interest
Concentration of phosphorylated Tau proteins in basal tears of patients with AD-dementia vs patients with AD-MCI | At inclusion
  12μL of tears will be collected using Schirmer strips after instillation of an anaesthetic eye drop. A multiplex analysis for the detection of protein of interest
Concentration of Amyloid β 1-40 proteins in basal tears of patients with AD-dementia vs patients with AD-MCI | At inclusion
  12μL of tears will be collected using Schirmer strips after instillation of an anaesthetic eye drop. A multiplex analysis for the detection of protein of interest
Concentration of Amyloid β 1-42 proteins in basal tears of patients with AD-dementia vs patients with AD-MCI | At inclusion
  12μL of tears will be collected using Schirmer strips after instillation of an anaesthetic eye drop. A multiplex analysis for the detection of protein of interest
Lipids in basal tears of patients with AD-dementia vs patients with AD-MCI | At inclusion
  Collection of tears (5μL) using a glass micropipette without local anaesthetic. Identification of lipids in basal tears using liquid chromatography-mass spectrometry.
Metabolites in basal tears of patients with AD-dementia vs patients with AD-MCI | At inclusion
  Collection of tears (5μL) using a glass micropipette without local anaesthetic. Identification of metabolites in basal tears using liquid chromatography-mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Victoire LEROY, MD, Study Director — CHRU de Tours
Locations (1):
- CHRU de Tours, Tours, France, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may obtain access to all deidentified data in COG-EYE on a substantial request.